CLINICAL TRIAL: NCT04885413
Title: An Open-label, Single Arm, Phase II Trial of Niraparib in Combination With Anti-PD1 Antibody in Recurrent/ Advanced Stage Endometrial Cancer Patients
Brief Title: An Open-label, Single Arm, Phase II Trial of Niraparib in Combination With Anti-PD1（Programmed Cell Death Protein 1） Antibody in Recurrent/ Advanced Stage Endometrial Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jundong Li, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SINI
Record Dates: First submitted 2021-05-11; First posted 2021-05-13 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Recurrent/ Advanced Stage Endometrial Cancer Patients
MeSH Terms: interventions — niraparib; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study arm (Experimental): Sintilimab： 200mg i.v., d1, 21days one cycle Niraparib： 200mg p.o qd，d1-d21, 21days one cycle
  Interventions: Drug: Niraparib in Combination With Anti-PD1 Antibody

INTERVENTIONS:
Drug: Niraparib in Combination With Anti-PD1 Antibody — Sintilimab： 200mg i.v., d1, 21days one cycle Niraparib： 200mg p.o qd，d1-d21, 21days one cycle
  Other Names: sintilimab

SUMMARY:
Endometrial carcinoma is the most common malignancy of the female reproductive tract. Most cases are diagnosed at an early stage due to the appearance of symptoms such as postmenopausal bleeding. However, endometrial carcinoma carries a poor prognosis when it recurs after previous definitive treatment or when diagnosed at an advanced stage.The 5-year survival rate for FIGO III is approximately 57-66% and for FIGO IV is approximately 10-20%.The combination of PARP（poly adenosine diphosphate-ribose polymerase）inhibitors and PD1/PD-L1 has the theoretical support of preclinical molecular biology. In recent years, a large number of basic studies and preclinical models have confirmed that this combination therapy has superimposed or even synergistic effects on multiple levels.This study intends to explore the efficacy and safety of anti-PD-1 antibody combined with niraparib in the treatment of recurrent or advanced endometrial cancer.

DETAILED DESCRIPTION:
This study is an open, multi-center, prospective single-arm Phase II study to study the effectiveness of niraparib combined with sintilimab in the treatment of recurrent/advanced endometrial cancer that has failed or cannot be tolerated by chemotherapy Sex and safety. The study intends to enroll 37 patients who have undergone histopathologically confirmed recurrence/advanced endometrial cancer who have experienced first-line and above chemotherapy failure or intolerance and received niraparib combined with sintilimab for treatment. The Simon two-stage design is used to estimate the sample size. For the first type of error, the value of α (one-sided) is 0.05, the value of β is 0.2, the test power is 0.8, and the ORR of the second-line chemotherapeutic drug is 15%. It is assumed that the objective population of niraparib combined with sintilimab in the treatment of the target subject population The remission rate was 35%. Nine cases were enrolled in the first stage. When the number of effective cases was ≤1, the combination therapy was considered to be no better than the single drug, and the trial was terminated. Otherwise, continue with the enrollment of 25 cases in the second stage. Assuming a loss rate of 10%, 37 subjects are expected to be enrolled in the trial.

ELIGIBILITY:
Inclusion Criteria:

1. The subject understands the trial process, signs an informed consent form, and agrees to participate in the research
2. 18-70 years of age and female;
3. Histologically confirmed endometrial epithelial carcinoma (including endometrioid adenocarcinoma, clear cell carcinoma, serous adenocarcinoma, dedifferentiated/undifferentiated endometrioid carcinoma), carcinosarcoma (excluding specific types of endometrial epithelial carcinoma such as small-cell neuroendocrine carcinoma), and excluding uterine sarcoma；
4. Recurrence or advanced endometrial cancer that is not suitable for local treatment. At least first-line chemotherapy has failed or is intolerant；Including the following

   * Patients with recurrent endometrial cancer have received at least first-line chemotherapy for recurrence, and imaging studies suggest disease progression during or after treatment
   * Advanced endometrial cancer (FIGO Stage III-IV) that has received neoadjuvant chemotherapy/adjuvant chemotherapy or radical concurrent radiotherapy and chemotherapy, disease progression during first-line chemotherapy or recurrence within 6 months of the end of first-line treatment
   * Patients with recurrent endometrial cancer cannot tolerate first-line chemotherapy
5. At least one measurable lesion by RECIST1.1 on CT;
6. Subjects provide formalin-fixed and paraffin-embedded tumor tissue samples for pathological consultation；
7. ECOG performance status 0-1;
8. Life expectancy ≥ 16 weeks;
9. Good organ function, including:

   * Neutrophil count ≥1500/µL (no growth factor support treatment within 7 days of the start of the study treatment)
   * Platelets ≥100,000/µL (Do not accept platelet transfusion and any form of platelet-increasing treatment within 2 weeks of the start of the study)
   * Hemoglobin ≥90g/L (transfusion should not be received within 2 weeks from the beginning of study treatment, and EPO should be required for support treatment within 7 days)
   * Serum creatinine ≤1.5 times the upper limit of normal, or creatinine clearance ≥60mL/min (according to the Cockcroft-Gault formula)
   * Total bilirubin ≤1.5 times the upper limit of normal or direct bilirubin ≤1.0 times the upper limit of normal
   * AST and ALT ≤2.5 times the upper limit of normal, liver metastasis must be ≤5 times the upper limit of normal
   * Urinary protein ≤ (+), or 24-hour urine protein quantification is less than 1g
   * Thyroid-stimulating hormone (TSH) ≤1xULN (if abnormal, also examine FT3, FT4, if normal, it can be included in the group)
   * Plasma cortisol ≤1xULN
   * International normalized ratio (INR) and activated partial thromboplastin time≤1.5ULN (unless anticoagulant therapy is being used due to disease)
10. The adverse effects of any previous treatment have returned to ≤CTCAE grade 1 or baseline, except for symptomatically stable sensory neuropathy or hair loss ≤CTCAE grade 2, except for anemia.
11. Previous hormonal or immunotherapy was permitted.
12. Women of reproductive age who had a negative pregnancy test at the time of enrolment and who committed to use adequate and effective contraception or abstinence for the period from the beginning to the end of the study and for a period of 3 months after the last administration of the study medication were eligible for enrolment

Exclusion Criteria:

1. Prior receipt of any PARP inhibitor;
2. Patients with other invasive cancers other than endometrial cancer within the first 5 years of enrollment, excluding complete treatment of various cancers in situ within 2 years, such as squamous cell skin cancer, breast cancer, etc.
3. The last systemic or radical antitumor therapy, including radiotherapy, chemotherapy, and targeted therapy (small molecule targeted therapy is within 2 weeks before the first administration), immunotherapy, and palliative radiation therapy for symptom control, was completed at least 2 weeks before the first administration.
4. Received Chinese patent medicines or Chinese herbal medicines or immunomodulatory drugs (thymus, interferon, interleukin, etc.) with anti-tumor effects 2 weeks before enrollment.
5. Have undergone major surgery within 4 weeks before the start of the study or are expected to undergo major surgery during the study period, or any surgical effects that have not yet recovered after the surgery.
6. Symptomatic, uncontrolled brain metastases or neumomeningeal metastases without the need for radiographic confirmation;Patients with spinal cord compression may still be considered if they received targeted treatment and have evidence of clinically stable > for at least 28 days (controlled CNS metastases must have been treated with treatment such as radiation or chemotherapy at least 1 month prior to study entry;Patients should not develop new symptoms associated with central nervous system lesions or symptoms indicative of disease progression, and patients should either take a steady dose of hormones or do not need hormones.)
7. Uncontrollable pleural and ascites.
8. Any active autoimmune disease or a history of autoimmune diseases (including but not limited to: autoimmune hepatitis, interstitial pneumonia, enteritis, hepatitis, nephritis, the pituitary gland inflammation, vasculitis, uveitis, or need to accept the system of sex hormone therapy and/or immunosuppressive therapy in patients with asthma (such as the need of bronchodilator), except the following:In the last 2 years without systematic treatment vitiligo, alopecia, Graves disease, psoriasis or eczema, stable immune thyroiditis controlled with treatment, type I diabetes requiring only stable insulin, childhood asthma has been completely remission.
9. Immunosuppressant or systemic hormonal therapy (>10mg/ d or other equivalent hormonal preparation) was being used for immunosuppressive purposes and continued to be used 2 weeks before enrollment. Topical and systemic use not exceeding >10mg/ d or other equivalent hormonal preparation was permitted.
10. With active bleeding (need) researchers to evaluate bleeding caused by tumor, with bleeding tendency or bleeding risk (such as tumor involving the great vessels, important bronchus, unable to control the obvious bleeding after hemostatic treatment, not cured bronchiectasis), or blood coagulation function apparently unusual, is treated with thrombolysis and anticoagulation (including need long-term antiplatelet therapy).
11. Thrombosis or embolism events in the past 6 months, such as cerebral vascular accident (including transient ischemic attack), pulmonary embolism;
12. Severe cardiovascular disease or medical history includes but not limited to the following:

    * NYHA (New York Heart Association) grade 3 and 4 congestive heart failure within 6 months before enrollment.
    * Suffered from unstable angina or newly diagnosed angina or myocardial infarction within 12 months before screening.
    * Arrhythmia requiring therapeutic intervention (Patients taking β-blockers or digoxin can be included in the group).
    * Valvular heart disease with CTCAE≥2.
    * Poorly controlled hypertension (systolic blood pressure> 150 mmHg or diastolic blood pressure> 100 mmHg;
13. Patients with moderate or above pulmonary dysfunction that cannot be relieved, interstitial pulmonary disease or active pulmonary tuberculosis;
14. Patients with active ulcers, intestinal perforation, unmitigated intestinal obstruction, and a history of gastrointestinal perforation during the 28 days prior to study enrollment.
15. Active inflammatory bowel disease, uncontrollable nausea and vomiting, inability to swallow study medication, any gastrointestinal disease that may interfere with drug absorption and metabolism;
16. Active infections such as human immunodeficiency virus, syphilis, untreated active hepatitis (HBV DNA copy number greater than 1000IU/ml, HCV RNA positive), etc.
17. Severe infection occurred 4 weeks before first administration;
18. Other serious or uncontrolled diseases.
19. Have received live vaccine or live attenuated vaccine 30 days before the first administration;
20. People who are known to be allergic to active or inactive ingredients of the study drug or a drug with a similar chemical structure;Patients who are pregnant or breastfeeding, or who are expected to become pregnant during the study treatment period;
21. Other laboratory abnormalities:

    * Uncorrectable hyponatremia (sodium <130 mmol/L; serum potassium <3.5 mmol/L);
    * Any prior or current disease, treatment, or laboratory abnormality that may interfere with the results of the study and affect the patient's full participation in the study, or that the investigator considers the patient unsuitable for participation in the study;
22. Any situation that the investigator deems unsuitable for participation, including poor understanding and coordination.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall respond rate | at 6 months
  The primary objective of this study is to determine the preliminary efficacy of administration of niraparib in combination with sintilimab in the treatment of recurrent/ advanced stage endometrial cancer, as measured by the objective response rate (ORR), which is a combination of CR (the target lesion completely disappeared over 4 weeks) and PR (Target lesions were reduced by more than 30% for more than 4 weeks).

SECONDARY OUTCOMES:
DoR（duration of response） | at 6 months
  From the start of Niraparib in Combination With sintilimab Antibody until progression or unacceptable toxicity.
PFS | 1 year
  Progression free survival
Overall survival rate | at 6 months
  Overall survival is defined as the time from registration to death from any cause, and subjects who are thought to be alive at the time of final analysis will be censored at the last date of contact.
Disease Control Rate | at 6 months
  The total proportion of subjects who have an objective tumor response (CR + PR+SD) using the RECIST criteria.
TTR | at 6 months
  Time to objective response
Adverse reaction rate | 30 days after completion of treatment
  As determined by CTCAE v5.0 in subjects with recurrent /advanced stage endometrial cancer receiving combination of niraparib and sintilimab

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Centre, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within six months after the trial complete
URL: http://www.medresman.org.cn